CLINICAL TRIAL: NCT01746108
Title: Immunogenicity, Safety and Reactogenicity Study of GSK Biologicals' Pneumococcal Vaccine (Synflorix™) When Administered to Children Who Are at an Increased Risk of Pneumococcal Infection
Brief Title: Immunogenicity and Safety Study of GlaxoSmithKline (GSK) Biologicals' Pneumococcal Vaccine (Synflorix™) When Administered to Children Who Are at an Increased Risk of Pneumococcal Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 115884; 2011-006013-34 (EudraCT Number)
Record Dates: First submitted 2012-11-28; First posted 2012-12-10 (Estimated); Results first posted 2017-01-09 (Estimated); Last update posted 2019-07-09 (Actual); Status verified 2019-06

CONDITIONS: Infections, Streptococcal; Streptococcus Pneumoniae Vaccines
Keywords: Pneumococcal infection; Synflorix; Children; Immunogenicity; Safety
MeSH Terms: conditions — Streptococcal Infections; Pneumococcal Infections | interventions — PHiD-CV vaccine

ARMS (4):
- At-risk-Unprimed Group (Experimental): Subjects who have not been previously vaccinated with any pneumococcal vaccine and are at an increased risk of pneumococcal infection.
  Interventions: Biological: Synflorix™
- At-risk-Primed Group (Experimental): Subjects who have been previously vaccinated
  * with at least one dose of a pneumococcal conjugate vaccine i.e. either Synflorix (10Pn-PD-DiT), Prevenar or Prevenar13.
  * with plain polysaccharide pneumococcal vaccine more than 2 years and less than 5 years before enrollment.
  and are at an increased risk of pneumococcal infection.
  Interventions: Biological: Synflorix™
- Healthy-Unprimed Group (Active Comparator): Subjects who have not been previously vaccinated with any pneumococcal vaccine and are healthy.
  Interventions: Biological: Synflorix™
- Healthy-Primed Group (Active Comparator): Subjects who have been previously vaccinated with at least one dose of a pneumococcal vaccine and are healthy.
  Interventions: Biological: Synflorix™

INTERVENTIONS:
Biological: Synflorix™ — 1 or 2 doses depending on the priming status, intramuscularly in the non-dominant deltoid muscle or the thigh.

SUMMARY:
The purpose of this study is to evaluate the immunogenicity, safety and reactogenicity of GSK Biologicals' 10Pn-PD-DiT vaccine in children aged between 2 and 17 years of age having asplenia, splenic dysfunction or complement deficiencies.

In addition, this study will include an age-matched control group of healthy children aged 24-59 months in order to descriptively compare the immunogenicity of 10Pn-PD-DiT vaccine in the at-risk population to that of the general, healthy population one month after each pneumococcal vaccination.

DETAILED DESCRIPTION:
The protocol has been amended to clarify the definition of priming status to consider for inclusion of subjects in the primed groups.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that parent(s)/Legally Acceptable Representative(s) [LAR(s)] can and will comply with the requirements of the protocol.
* Written informed consent obtained from the parent(s)/LAR(s) of the subject and informed assent obtained from the subject, if appropriate, prior to enrollment.
* Female subjects of non-child bearing potential may be enrolled in the study. (Non-child bearing potential is defined as pre-menarche, current tubal ligation, hysterectomy or ovariectomy).
* Female subjects of child bearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to the first vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Priming status:

* Children who have not been previously vaccinated with any pneumococcal vaccine, i.e. either plain polysaccharide pneumococcal vaccine, Synflorix (10Pn-PD-DiT), Prevenar or Prevenar13 will be considered for inclusion in the unprimed groups.

Children who have been previously vaccinated with:

* at least one dose of a pneumococcal conjugate vaccine, i.e. either Synflorix (10Pn-PD-DiT), Prevenar or Prevenar13
* with plain polysaccharide pneumococcal vaccine more than 2 years and less than 5 years before enrollment.
* will be considered for inclusion in the primed groups.

Additional inclusion criteria for the At-risk groups:

* A male or female aged between, and including, 2 and 17 years at the time of first vaccination.
* For the purpose of this study, at-risk subject is a subject with:

  * Congenital or acquired asplenia such as anatomic, surgical or functional asplenia or
  * Splenic dysfunction, chronic gastrointestinal disorders, liver disease, infiltrative disorders, vascular disorder etc or

Note: All individuals who are diagnosed by the investigator as with splenic dysfunction are eligible for enrollment in the At-risk group. When available, investigator will collect medical documentation for reduced splenic function diagnosed with an appropriate technique in the At-risk subject's medical records. No further assessment will be necessary. A maximum of 35 individuals with sickle-cell disease can be enrolled in the At-risk group. These subjects do not require assessment of the splenic function as sickle-cell disease is invariably associated with severe splenic dysfunction.

- Complement deficiencies. For all subjects defined as At-risk the Investigator will make all efforts to collect information from the subject/subject's parent(s)/LAR(s) during the interview and/or from previously available medical documentation on the date and conditions which have made a child at-risk of pneumococcal infection and/or the results of tests determining spleen dysfunction or complement deficiency. This should be documented in the medical records of the At-risk subject. No originals/copies of medical documentation are needed.

Additional inclusion criteria for the Healthy group:

* A male or female matched (for age and country) to a subject aged 24-59 months from the At-risk group.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol during the period starting 30 days before each dose of vaccine(s) and ending 30 days after*.

  * In case an emergency mass vaccination for an unforeseen public health threat is organised by the public health authorities, outside the routine immunization program, vaccines can be administered at any time during the study period provided it is licensed and used according to its Summary of Product Characteristics or Prescribing Information and according to the local governmental recommendations and that a written approval of the Sponsor is provided. Vaccines that are recommended for subjects with an increased risk of bacterial infection, can be administered at any time to the subjects enrolled in the At-risk group.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* History of any neurological disorders or seizures.
* Acute disease and/or fever at the time of enrollment.
* History of chronic alcohol consumption and/or drug abuse.
* Any confirmed or suspected Human Immunodeficiency virus (HIV) infection, based on medical history and physical examination.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Major congenital defects except medical conditions that define an At-risk subject.
* Previous vaccination against pneumococcal infection with pneumococcal conjugate vaccine within the last 8 weeks.
* Previous vaccination against pneumococcal infection with plain polysaccharide vaccine within the last 2 years.

Additional exclusion criteria for the Healthy group:

* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose. Inhaled and topical steroids are allowed.
* Serious chronic illness.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Family history of congenital or hereditary immunodeficiency.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2013-06-18 (Actual); Primary Completion 2015-06-29 (Actual); Study Completion 2015-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- Poland (3):
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
- Russia (3):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Novokuznetsk
  - GSK Investigational Site, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Background] Szenborn L, Osipova IV, Czajka H, Kharit SM, Jackowska T, Francois N, Habib MA, Borys D. Immunogenicity, safety and reactogenicity of the pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) in 2-17-year-old children with asplenia or splenic dysfunction: A phase 3 study. Vaccine. 2017 Sep 25;35(40):5331-5338. doi: 10.1016/j.vaccine.2017.08.039. Epub 2017 Aug 31. PMID 28866290
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: No healthy primed subjects were enrolled in the study.
Groups:
- Synflorix AR-Pr-2-17Y Group: Primed (Pr) subjects aged between 24 months and 17 years, who were at an increased risk (AR) of pneumococcal infection*, receiving 1 dose of SynflorixTM vaccine: Primed groups included subjects who have been previously vaccinated with at least one dose of a pneumococcal conjugate vaccine, i.e. either SynflorixTM, PrevenarTM or Prevenar13TM or with plain polysaccharide pneumococcal vaccine more than 2 years (24 months) and less than 5 years (60 months) before enrolment.
  *An at-risk subject was a subject with Congenital or acquired asplenia such as anatomic, surgical or functional asplenia, or Splenic dysfunction [some degree of functional asplenia, such as sickle-cell disease and other hemoglobinopathies, Hodgkin disease, rheumatologic diseases, systemic lupus erythematous (SLE), chronic gastrointestinal disorders, liver disease, infiltrative disorders, vascular disorder etc.] or Complement deficiencies, e.g.C1-C4, C5-C9, properdin factor H or factor D.
- Synflorix AR-Un-2-17Y Group: Unprimed (Un) subjects aged between 24 months and 17 years, who were at an increased risk (AR) of pneumococcal infection*, receiving 2 doses of SynflorixTM vaccine: Unprimed groups included subjects who have not been previously vaccinated with any pneumococcal vaccine, i.e. either plain polysaccharide pneumococcal vaccine, SynflorixTM, PrevenarTM or Prevenar13TM.
  *An at-risk subject was a subject with Congenital or acquired asplenia such as anatomic, surgical or functional asplenia, or Splenic dysfunction [some degree of functional asplenia, such as sickle-cell disease and other hemoglobinopathies, Hodgkin disease, rheumatologic diseases, systemic lupus erythematous (SLE), chronic gastrointestinal disorders, liver disease, infiltrative disorders, vascular disorder etc.] or Complement deficiencies, e.g.C1-C4, C5-C9, properdin factor H or factor D.
- Synflorix HE-Un-2-4Y Group: Healthy (HE) unprimed (Un) subjects, aged between 24 and 59 months of age (age-matched to the subjects aged 24-59 months in the At risk groups), receiving 2 doses of SynflorixTM vaccine. Unprimed groups included subjects who have not been previously vaccinated with any pneumococcal vaccine, i.e. either plain polysaccharide pneumococcal vaccine, SynflorixTM, PrevenarTM or Prevenar13TM. For each enrolled at-risk subject aged between 24-59 months, a healthy subject of the same age expressed in years from the same country should be enrolled regardless of the priming status (i.e.: a healthy subject could be enrolled only once if he/she could be matched with an unmatched at-risk subject of the same age and country).
Period: Overall Study
Arm/Group | Synflorix AR-Pr-2-17Y Group | Synflorix AR-Un-2-17Y Group | Synflorix HE-Un-2-4Y Group
Started | 18 | 28 | 6
Completed | 18 | 24 | 6
Not Completed | 0 | 4 | 0
Not completed — Migrated /moved from study area | 0 | 1 | 0
Not completed — Adverse event, non-fatal | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Synflorix AR-Pr-2-17Y Group | Synflorix AR-Un-2-17Y Group | Synflorix HE-Un-2-4Y Group | Total
Number analyzed (Participants) | 18 | 28 | 6 | 52
Age, Continuous [Mean (Standard Deviation); unit: Years] | 11.3 (3.8) | 8.6 (4.2) | 2.8 (0.8) | 8.87 (4.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 2 | 26
  Male | 8 | 14 | 4 | 26

OUTCOME MEASURES:

1. Primary Outcome: Concentrations of Antibodies Against Vaccine Pneumococcal Serotypes in the At Risk Primed Group.
Description: Antibodies assessed for this outcome measure were those against the vaccine pneumococcal serotypes 1, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F (ANTI-1, -4, -5, -6A, -6B, -7F, -9V, -14, -18C, -19A, -19F and -23F). Antibody concentrations were measured by 22F-inhibition enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per millilitre (μg/mL). The seropositivity cut-off of the assay was an antibody concentration ≥ 0.05 μg/mL.
  Antibody concentrations < 0.05 μg/mL were given an arbitrary value of half the cut-off for the purpose of GMC calculation.
Time Frame: One month after Dose 1 (At Month 1)
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom assay results were available for antibodies against at least one pneumococcal vaccine serotype or protein D for at least one blood sample taken after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix AR-Pr-2-17Y Group
Number analyzed (Participants) | 18
μg/mL
  Anti-1 (N=18) | 1.94 [1.4 to 2.69]
  Anti-4 (N=18) | 6.16 [3.89 to 9.76]
  Anti-5 (N=18) | 2.44 [1.24 to 4.83]
  Anti-6B (N=18) | 3.66 [1.93 to 6.96]
  Anti-7F (N=18) | 3.34 [2.54 to 4.38]
  Anti-9V (N=18) | 2.87 [1.65 to 4.97]
  Anti-14 (N=18) | 21.08 [10.97 to 40.52]
  Anti-18C (N=18) | 10.84 [6.99 to 16.81]
  Anti-19F (N=18) | 18.22 [9.57 to 34.7]
  Anti-23F (N=18) | 2.24 [1.14 to 4.41]
  Anti-6A (N=18) | 3.76 [1.7 to 8.34]
  Anti-19A (N=18) | 4.44 [2.34 to 8.45]

2. Primary Outcome: Concentrations of Antibodies Against Vaccine Pneumococcal Serotypes in the At Risk Un-primed Group.
Description: as for outcome 1
Time Frame: One month after Dose 1 (At Month 1) and one month after Dose 2 (At Month 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix AR-Un-2-17Y Group
Number analyzed (Participants) | 23
μg/mL
  Anti-1 Month 1 (N=23) | 1.52 [1.13 to 2.06]
  Anti-1 Month 3 (N=21) | 2.52 [1.87 to 3.4]
  Anti-4 Month 1 (N=23) | 9.26 [6.62 to 12.95]
  Anti-4 Month 3 (N=21) | 7.67 [5.59 to 10.53]
  Anti-5 Month 1 (N=23) | 2.74 [1.6 to 4.69]
  Anti-5 Month 3 (N=21) | 3.93 [2.46 to 6.27]
  Anti-6B Month 1 (N=23) | 1.21 [0.59 to 2.46]
  Anti-6B Month 3 (N=21) | 2.19 [1.26 to 3.8]
  Anti-7F Month 1 (N=23) | 3.25 [2.24 to 4.71]
  Anti-7F Month 3 (N=21) | 5.6 [3.95 to 7.93]
  Anti-9V Month 1 (N=23) | 1.89 [1.14 to 3.12]
  Anti-9V Month 3 (N=21) | 3.23 [2.07 to 5.03]
  Anti-14 Month 1 (N=23) | 7.78 [3.86 to 15.68]
  Anti-14 Month 3 (N=21) | 13.64 [8.42 to 22.12]
  Anti-18C Month 1 (N=23) | 13.04 [8.08 to 21.04]
  Anti-18C Month 3 (N=21) | 24.15 [15.4 to 37.86]
  Anti-19F Month 1 (N=23) | 12.41 [6.05 to 25.44]
  Anti-19F Month 3 (N=21) | 20.53 [11.42 to 36.9]
  Anti-23F Month 1 (N=23) | 1.09 [0.5 to 2.4]
  Anti-23F Month 3 (N=21) | 2.26 [1.27 to 4.04]
  Anti-6A Month 1 (N=23) | 1.02 [0.53 to 1.97]
  Anti-6A Month 3 (N=21) | 1.5 [0.87 to 2.58]
  Anti-19A Month 1 (N=23) | 2.18 [0.96 to 4.95]
  Anti-19A Month 3 (N=21) | 4.05 [1.96 to 8.38]

3. Primary Outcome: Opsonophagocytic Titers Against Vaccine Pneumococcal Serotypes in the At Risk Primed Group.
Description: Pneumococcal vaccine serotypes assessed were 1, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F and were calculated, expressed as geometric mean titers (GMTs). The seropositivity cut-off for the assay was
  ≥ 8. Antibody titers < 8 were given an arbitrary value of half the cut-off for the purpose of GMT calculation.
Time Frame: One month after Dose 1 (At Month 1)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix AR-Pr-2-17Y Group
Number analyzed (Participants) | 15
Titers
  Opsono-1 (N=14) | 12.4 [5.3 to 29.3]
  Opsono-4 (N=15) | 1291.6 [722.5 to 2308.9]
  Opsono-5 (N=15) | 75.9 [26.9 to 214.2]
  Opsono-6B (N=15) | 698.1 [348.8 to 1397.2]
  Opsono-7F (N=15) | 2787.4 [1959.9 to 3964.4]
  Opsono-9V (N=15) | 1955.3 [1209.8 to 3160.3]
  Opsono-14 (N=15) | 2495.7 [1220.6 to 5103.1]
  Opsono-18C (N=15) | 4421.4 [2982.8 to 6553.9]
  Opsono-19F (N=15) | 3272.4 [1849.4 to 5790.5]
  Opsono-23F (N=15) | 613.8 [244.9 to 1538.5]
  Opsono-6A (N=15) | 2590.9 [1394.2 to 4814.7]
  Opsono-19A (N=15) | 961.2 [376.4 to 2454.8]

4. Primary Outcome: Opsonophagocytic Titers Against Vaccine Pneumococcal Serotypes in the At Risk Un-primed Group.
Description: as for outcome 3
Time Frame: One month after Dose 1 (At Month 1) and one month after Dose 2 (At Month 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix AR-Un-2-17Y Group
Number analyzed (Participants) | 17
Titers
  Opsono-1 Month 1 (N=14) | 8.6 [4 to 18.6]
  Opsono-1 Month 3 (N=15) | 29.1 [12.1 to 70.1]
  Opsono-4 Month 1 (N=17) | 1497.1 [696.6 to 3217.4]
  Opsono-4 Month 3 (N=16) | 2657 [1763.5 to 4003.3]
  Opsono-5 Month 1 (N=16) | 112.5 [49.1 to 258]
  Opsono-5 Month 3 (N=16) | 212.9 [116 to 390.7]
  Opsono-6B Month 1 (N=16) | 1188.8 [548.7 to 2575.7]
  Opsono-6B Month 3 (N=16) | 2384.3 [1483.2 to 3832.8]
  Opsono-7F Month 1 (N=17) | 4433.6 [3110.8 to 6319]
  Opsono-7F Month 3 (N=16) | 6724.3 [4240.9 to 10661.8]
  Opsono-9V Month 1 (N=17) | 1076.5 [330.8 to 3502.8]
  Opsono-9V Month 3 (N=16) | 1319.5 [677.2 to 2571.1]
  Opsono-14 Month 1 (N=17) | 2724.6 [1473.1 to 5039.1]
  Opsono-14 Month 3 (N=16) | 6590.5 [3329.7 to 13044.6]
  Opsono-18C Month 1 (N=17) | 8665.8 [5076.4 to 14793.2]
  Opsono-18C Month 3 (N=16) | 9939.8 [7045 to 14024.1]
  Opsono-19F Month 1 (N=16) | 4569.1 [2695.3 to 7745.5]
  Opsono-19F Month 3 (N=16) | 3441.8 [1709.8 to 6928]
  Opsono-23F Month 1 (N=16) | 1326.4 [796.1 to 2210]
  Opsono-23F Month 3 (N=16) | 1949.3 [1145.5 to 3317.2]
  Opsono-6A Month 1 (N=16) | 1982.6 [648.9 to 6057.2]
  Opsono-6A Month 3 (N=14) | 1908.3 [975.1 to 3734.8]
  Opsono-19A Month 1 (N=16) | 1037.4 [373.5 to 2881.5]
  Opsono-19A Month 3 (N=16) | 2769.3 [1490.6 to 5145]

5. Primary Outcome: Concentrations of Antibodies Against Protein D (PD) in the At Risk Primed Group.
Description: Anti-protein D (Anti-PD) antibody concentrations by Enzyme-Linked Immunosorbent Assay (ELISA) were calculated, expressed as geometric mean concentrations (GMCs) in ELISA unit per millilitre (EL.U/mL) and tabulated. The seropositivity cut-off for the assay was ≥ 153 EL.U/mL. Antibody concentrations < 153 EL.U/mL were given an arbitrary value of half the cut-off for the purpose of GMC calculation.
Time Frame: One month after Dose 1 (At Month 1)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix AR-Pr-2-17Y Group
Number analyzed (Participants) | 18
EL.U/mL | 173.1 [109.2 to 274.3]

6. Primary Outcome: Concentrations of Antibodies Against Protein D (PD) in the At Risk Unprimed Group.
Description: as for outcome 5
Time Frame: One month after Dose 1 (At Month 1) and one month after Dose 2 (At Month 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix AR-Un-2-17Y Group
Number analyzed (Participants) | 23
EL.U/mL
  Anti-PD Month 1 (N=23) | 372.5 [179.3 to 773.8]
  Anti-PD Month 3 (N=19) | 870.8 [420.6 to 1803]

7. Secondary Outcome: Number of Subjects With Any and Severe (Grade 3) Solicited Local Adverse Events (AEs) After Dose 1 for Subjects Aged Between 2 to 4 Years.
Description: Solicited local AEs assessed were pain, redness and swelling. Any = incidence of any local symptom regardless of intensity grade. Grade 3 pain = cried when limb was moved/spontaneously painful. Grade 3 redness/swelling = redness/swelling above 30 millimetre. Primed subjects received one dose and Unprimed subjects received two doses.
Time Frame: During the 4-day (Days 0-3) after dose 1
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Number; unit: Subjects
Groups:
- Synflorix AR-PR-2-4Y Group: Subset of the AR-PR-2-17Y Group including subjects aged between 24 and 59 months.
- Synflorix AR-Un-2-4Y Group: Subset of the AR-UN-2-17Y Group including subjects aged between 24 and 59 months.
Arm/Group | Synflorix HE-Un-2-4Y Group | Synflorix AR-PR-2-4Y Group | Synflorix AR-Un-2-4Y Group
Number analyzed (Participants) | 6 | 1 | 5
Subjects
  Any pain Dose 1 | 5 | 1 | 2
  Grade 3 pain Dose 1 | 1 | 0 | 0
  Any redness Dose 1 | 6 | 1 | 2
  Grade 3 redness Dose 1 | 2 | 0 | 0
  Any swelling Dose 1 | 3 | 1 | 1
  Grade 3 Swelling Dose 1 | 1 | 0 | 1

8. Secondary Outcome: Number of Subjects With Any and Severe (Grade 3) Solicited Local Adverse Events (AEs) After Dose 2 for Subjects Aged Between 2 to 4 Years.
Description: as for outcome 7
Time Frame: During the 4-day (Days 0-3) after dose 2
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Synflorix HE-Un-2-4Y Group | Synflorix AR-Un-2-4Y Group
Number analyzed (Participants) | 6 | 2
Subjects
  Any pain Dose 2 | 3 | 1
  Grade 3 pain Dose 2 | 1 | 0
  Any redness Dose 2 | 4 | 0
  Grade 3 Redness Dose 2 | 0 | 0
  Any swelling Dose 2 | 1 | 1
  Grade 3 Swelling Dose 2 | 0 | 0

9. Secondary Outcome: Number of Subjects With Any and Severe (Grade 3) Solicited Local Adverse Events (AEs) After Dose 1 for Subjects Aged Between 5 to 17 Years.
Description: Solicited local AEs assessed were pain, redness and swelling. Any = incidence of any local symptom regardless of intensity grade. Grade 3 pain =Significant pain at rest. Prevented normal every day activities. Grade 3 redness/swelling = redness/swelling above 50 millimetre. Primed subjects received one dose and Unprimed subjects received two doses.
Time Frame: During the 4-day (Days 0-3) after dose 1
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Number; unit: Subjects
Groups:
- Synflorix AR-PR-5-17Y Group: Subset of the AR-PR-2-17Y Group including subjects aged between 5 and 17 years.
- Synflorix AR- UN-5-17Y Group: Subset of the AR- UN-5-17Y Group including subjects aged between 5 and 17 years.
Arm/Group | Synflorix AR-PR-5-17Y Group | Synflorix AR- UN-5-17Y Group
Number analyzed (Participants) | 17 | 23
Subjects
  Any pain Dose 1 | 14 | 22
  Grade 3 pain Dose 1 | 0 | 4
  Any redness Dose 1 | 6 | 10
  Grade 3 redness Dose 1 | 0 | 0
  Any swelling Dose 1 | 4 | 6
  Grade 3 Swelling Dose 1 | 1 | 0

10. Secondary Outcome: Number of Subjects With Any and Severe (Grade 3) Solicited Local Adverse Events (AEs) After Dose 2 for Subjects Aged Between 5 to 17 Years.
Description: Solicited local AEs assessed were pain, redness and swelling. Any = incidence of any local symptom regardless of intensity grade. Grade 3 pain = Significant pain at rest. Prevented normal every day activities. Grade 3 redness/swelling = redness/swelling above 50 millimetre. Primed subjects received one dose and Unprimed subjects received two doses.
Time Frame: During the 4-day (Days 0-3) after dose 2
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Synflorix AR- UN-5-17Y Group
Number analyzed (Participants) | 23
Subjects
  Any pain Dose 2 | 16
  Grade 3 pain Dose 2 | 1
  Any redness Dose 2 | 7
  Grade 3 redness Dose 2 | 1
  Any swelling Dose 2 | 5
  Grade 3 Swelling Dose 2 | 3

11. Secondary Outcome: Number of Subjects With Any, Severe (Grade 3) and Related Solicited General Adverse Events (AEs) After Dose 1 for Subjects Aged Between 2 to 4 Years.
Description: General AEs = drowsiness, irritability, loss of appetite (loss of appet) and fever (axillary ≥ 37.5 degrees Celsius). Any= Incidence of any solicited general symptom regardless of intensity grade or relationship to vaccination. Grade 3: drowsiness = prevented normal activity; irritability = crying that could not be comforted/ prevented normal activity; loss of appetite = not eating at all; fever > 39.5°C. Related = symptom assessed by the investigator as related to the vaccination. Primed subjects received one dose and Unprimed subjects received two doses.
Time Frame: During the 4-day (Days 0-3) after dose 1
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Synflorix HE-Un-2-4Y Group | Synflorix AR-PR-2-4Y Group | Synflorix AR-Un-2-4Y Group
Number analyzed (Participants) | 6 | 1 | 5
Subjects
  Any drowsiness Dose 1 | 1 | 1 | 0
  Grade 3 drowsiness Dose 1 | 0 | 0 | 0
  Related drowsiness Dose 1 | 1 | 1 | 0
  Any irritability Dose 1 | 3 | 1 | 1
  Grade 3 irritability Dose 1 | 0 | 0 | 0
  Related irritability Dose 1 | 3 | 1 | 1
  Any loss of appet Dose 1 | 4 | 1 | 2
  Grade 3 loss of appet. Dose 1 | 0 | 0 | 0
  Related loss of appet. Dose 1 | 3 | 1 | 1
  Any Fever Dose 1 | 1 | 0 | 1
  Grade 3 Fever Dose 1 | 0 | 0 | 0
  Related fever Dose 1 | 1 | 0 | 0

12. Secondary Outcome: Number of Subjects With Any, Severe (Grade 3) and Related Solicited General Adverse Events (AEs) After Dose 2 for Subjects Aged Between 2 to 4 Years.
Description: as for outcome 11
Time Frame: During the 4-day (Days 0-3) after dose 2
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Synflorix HE-Un-2-4Y Group | Synflorix AR-Un-2-4Y Group
Number analyzed (Participants) | 6 | 2
Subjects
  Any drowsiness Dose 2 | 1 | 1
  Grade 3 drowsiness Dose 2 | 0 | 0
  Related drowsiness Dose 2 | 1 | 1
  Any irritability Dose 2 | 1 | 1
  Grade 3 irritability Dose 2 | 0 | 0
  Related irritability Dose 2 | 1 | 1
  Any loss of appet Dose 2 | 2 | 1
  Grade 3 loss of appet. Dose 2 | 0 | 0
  Related loss of appet. Dose 2 | 2 | 1
  Any Fever Dose 2 | 0 | 1
  Grade 3 Fever Dose 2 | 0 | 0
  Related fever Dose 2 | 0 | 1

13. Secondary Outcome: Number of Subjects With Any, Severe (Grade 3) and Related Solicited General Adverse Events (AEs) After Dose 1 for Subjects Aged Between 5 to 17 Years.
Description: General AEs = headache, fatigue, gastrointestinal symptoms (gastro symp) (nausea, vomiting, diarrhoea and/or abdominal pain) and fever (axillary ≥ 37.5 degrees Celsius). Any= Incidence of any solicited general symptom regardless of intensity grade or relationship to vaccination. Grade 3: headache, fatigue and gastrointestinal symptoms = symptoms that prevented normal activity; Fever > 39.5°C. Related = symptom assessed by the investigator as related to the vaccination. Primed subjects received one dose and Unprimed subjects received two doses.
Time Frame: During the 4-day (Days 0-3) after dose 1
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Synflorix AR-PR-5-17Y Group | Synflorix AR- UN-5-17Y Group
Number analyzed (Participants) | 17 | 23
Subjects
  Any fatigue Dose 1 | 5 | 5
  Grade 3 fatigue Dose 1 | 0 | 0
  Related fatigue Dose 1 | 4 | 4
  Any gastro symp Dose 1 | 3 | 4
  Grade 3 gastro symp. Dose 1 | 0 | 0
  Related gastro symp. Dose 1 | 2 | 0
  Any headache Dose 1 | 5 | 6
  Grade 3 headache Dose 1 | 0 | 0
  Related headache Dose 1 | 5 | 6
  Any Fever Dose 1 | 0 | 2
  Grade 3 Fever Dose 1 | 0 | 0
  Related fever Dose 1 | 0 | 2

14. Secondary Outcome: Number of Subjects With Any, Severe (Grade 3) and Related Solicited General Adverse Events (AEs) After Dose 2 for Subjects Aged Between 5 to 17 Years.
Description: as for outcome 13
Time Frame: During the 4-day (Days 0-3) after dose 2
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Synflorix AR- UN-5-17Y Group
Number analyzed (Participants) | 23
Subjects
  Any fatigue Dose 2 | 7
  Grade 3 fatigue Dose 2 | 0
  Related fatigue Dose 2 | 6
  Any gastro symp Dose 2 | 2
  Grade 3 gastro symp. Dose 2 | 0
  Related gastro symp. Dose 2 | 0
  Any headache Dose 2 | 5
  Grade 3 headache Dose 2 | 0
  Related headache Dose 2 | 5
  Any Fever Dose 2 | 1
  Grade 3 Fever Dose 2 | 0
  Related fever Dose 2 | 1

15. Secondary Outcome: Number of Subjects With Unsolicited AEs.
Description: An unsolicited adverse event is any adverse event (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: Within the 31-day (Days 0-30) post- vaccination period
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Synflorix AR-Pr-2-17Y Group | Synflorix AR-Un-2-17Y Group | Synflorix HE-Un-2-4Y Group
Number analyzed (Participants) | 18 | 28 | 6
Subjects | 2 | 14 | 4

16. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs).
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of study subjects
Time Frame: From Dose 1 at Month 0 up to study end at Month 1 for primed subjects and at Month 3 for unprimed subjects.
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Synflorix AR-Pr-2-17Y Group | Synflorix AR-Un-2-17Y Group | Synflorix HE-Un-2-4Y Group
Number analyzed (Participants) | 18 | 28 | 6
Subjects | 0 | 1 | 0

17. Secondary Outcome: Concentrations of Antibodies Against Vaccine Pneumococcal Serotypes in the Healthy Un-primed Group.
Description: as for outcome 1
Time Frame: One month after Dose 1 (At Month 1) and one month after Dose 2 (At Month 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix HE-Un-2-4Y Group
Number analyzed (Participants) | 4
EL.U/mL
  Anti-1 Month 1 (N=2) | 6.09 [0 to 90592008]
  Anti-1 Month 3 (N=4) | 2.41 [0.23 to 25.58]
  Anti-4 Month 1 (N=2) | 10.68 [0.03 to 4390.15]
  Anti-4 Month 3 (N=4) | 10.89 [6.53 to 18.18]
  Anti-5 Month 1 (N=2) | 2.29 [0.62 to 8.41]
  Anti-5 Month 3 (N=4) | 3 [1.2 to 7.53]
  Anti-6B Month 1 (N=3) | 0.52 [0.02 to 16.94]
  Anti-6B Month 3 (N=4) | 0.95 [0.29 to 3.14]
  Anti-7F Month 1 (N=3) | 7.62 [3.05 to 19.01]
  Anti-7F Month 3 (N=4) | 8.4 [2.98 to 23.71]
  Anti-9V Month 1 (N=3) | 2.51 [0.32 to 19.96]
  Anti-9V Month 3 (N=4) | 2.78 [0.77 to 10.01]
  Anti-14 Month 1 (N=2) | 1.44 [0.24 to 8.73]
  Anti-14 Month 3 (N=4) | 7.44 [5.12 to 10.81]
  Anti-18C Month 1 (N=3) | 7.36 [1.99 to 27.26]
  Anti-18C Month 3 (N=4) | 13.72 [2.57 to 73.26]
  Anti-19F Month 1 (N=2) | 20.23 [0.28 to 1466.83]
  Anti-19F Month 3 (N=4) | 12.87 [2.69 to 61.53]
  Anti-23F Month 1 (N=2) | 1.13 [0 to 1209.69]
  Anti-23F Month 3 (N=4) | 1.99 [0.37 to 10.63]
  Anti-6A Month 1 (N=2) | 0.89 [0 to 25368671]
  Anti-6A Month 3 (N=4) | 0.78 [0.26 to 2.29]
  Anti-19A Month 1 (N=2) | 0.1 [0 to 8.09]
  Anti-19A Month 3 (N=4) | 0.53 [0.16 to 1.74]

18. Secondary Outcome: Opsonophagocytic Titers Against Vaccine Pneumococcal Serotypes in the Healthy Un-primed Group.
Description: Pneumococcal vaccine serotypes assessed were 1, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F and were calculated, expressed as geometric mean titers (GMTs). The seropositivity cut-off for the assay was ≥ 8. Antibody titers < 8 were given an arbitrary value of half the cut-off for the purpose of GMT calculation. When number of subjects analysed = 1, Lower limit and Upper Limit values were entered as equal to the Geometric mean value. "999999.9" was used as placeholder when Upper Limit value was greater than "1.0E8".
Time Frame: One month after Dose 1 (At Month 1) and/or one month after Dose 2 (At Month 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix HE-Un-2-4Y Group
Number analyzed (Participants) | 2
Titers
  Opsono-1 Month 1 (N=2) | 35.2 [0 to 999999.9]
  Opsono-1 Month 3 (N=2) | 31.5 [0 to 999999.9]
  Opsono-4 Month 1 (N=2) | 1716.7 [556.1 to 5299.7]
  Opsono-4 Month 3 (N=2) | 3780.1 [0.2 to 62503343]
  Opsono-5 Month 3 (N=2) | 113.3 [0.2 to 61692.5]
  Opsono-6B Month 1 (N=2) | 891.3 [22.4 to 35452]
  Opsono-6B Month 3 (N=2) | 1118.1 [2.3 to 534561.1]
  Opsono-7F Month 1 (N=2) | 4789.2 [28.3 to 810373.3]
  Opsono-7F Month 3 (N=2) | 5269.9 [401.1 to 69232.8]
  Opsono-9V Month 1 (N=2) | 1121 [93.6 to 13432.2]
  Opsono-9V Month 3 (N=2) | 2999.8 [82.6 to 108968.9]
  Opsono-14 Month 1 (N=2) | 1344.9 [0.3 to 5396843]
  Opsono-14 Month 3 (N=2) | 7678.4 [3059.7 to 19269.1]
  Opsono-18C Month 1 (N=2) | 4462 [0.2 to 999999.9]
  Opsono-18C Month 3 (N=2) | 6269.6 [1176.4 to 33412.6]
  Opsono-19F Month 1 (N=2) | 1934.7 [506.3 to 7392.9]
  Opsono-19F Month 3 (N=2) | 1970.4 [250.1 to 15523.1]
  Opsono-23F Month 1 (N=2) | 420.6 [2 to 88878.1]
  Opsono-23F Month 3 (N=2) | 1324.5 [131 to 13391.2]
  Opsono-6A Month 1 (N=2) | 188.8 [0 to 999999.9]
  Opsono-6A Month 3 (N=2) | 2182.1 [1713.7 to 2778.5]
  Opsono-19A Month 1 (N=1) | 4 [4 to 4]
  Opsono-19A Month 3 (N=2) | 637.1 [35.9 to 11317.6]

19. Secondary Outcome: Concentrations of Antibodies Against Protein D (PD) in the Healthy Unprimed Group.
Description: as for outcome 5
Time Frame: One month after Dose 1 (At Month 1) and one month after Dose 2 (At Month 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix HE-Un-2-4Y Group
Number analyzed (Participants) | 4
EL.U/mL
  Anti-PD Month 1 (N=2) | 217.8 [35.9 to 1320.8]
  Anti-PD Month 3 (N=4) | 373.9 [140.1 to 998.3]

ADVERSE EVENTS:
Time Frame: SAEs: from Month 0 up to Study end, Solicited and Unsolicited AEs: within the 31-day post- vaccination period.
Arm/Group | Synflorix AR-Pr-2-17Y Group | Synflorix HE-Un-2-4Y Group | Synflorix AR-Un-2-17Y Group
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/6 | 1/28
Other Adverse Events (participants affected / at risk) | 17/18 | 6/6 | 27/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Synflorix AR-Pr-2-17Y Group (N=18) | Synflorix HE-Un-2-4Y Group (N=6) | Synflorix AR-Un-2-17Y Group (N=28)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Synflorix AR-Pr-2-17Y Group (N=18) | Synflorix HE-Un-2-4Y Group (N=6) | Synflorix AR-Un-2-17Y Group (N=28)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 5 (5) | 0 (0) | 7 (11)
Somnolence (Nervous system disorders) | 1 (1) | 1 (2) | 3 (3)
Fatigue (General disorders) | 5 (5) | 0 (0) | 10 (12)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 15 (15) | 5 (8) | 24 (41)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 4 (5)
Swelling (General disorders) | 5 (5) | 3 (4) | 10 (13)
Irritability (Psychiatric disorders) | 1 (1) | 4 (4) | 1 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 3 (3) | 0 (0) | 5 (6)
Erythema (Skin and subcutaneous tissue disorders) | 7 (7) | 6 (10) | 12 (19)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 4 (6) | 2 (3)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.